CLINICAL TRIAL: NCT04636099
Title: Preoperative CTA to Evaluate the Influence of Gastric Artery Type on the Clinical Outcome of Gastric Cancer Patients With BMI≥25.0 kg/m2：A Multicenter Randomized Controlled Study
Brief Title: Gastrointestinal Surgery Study Group 2001
Acronym: GISSG2001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: Qilu Hospital of Shandong University (Other); Shandong Provincial Hospital (Other Government); Qianfoshan Hospital (Other); Yantai Yuhuangding Hospital (Other); Weifang Medical University (Other); Weifang People's Hospital (Other); Jining First People's Hospital (Other); Weihai Municipal Hospital (Other); Weihai Central Hospital (Other); Dongying People's Hospital (Other); Rizhao People's Hospital (Other); People's Hospital of Jimo District, Qingdao (Unknown); Liaocheng People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QYFYKYLL791311920
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Gastrostomy; Computed Tomography Angiography; Clinical Outcome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTA Group (Experimental): The CTA group was peformed upper abdomen enhenced and CT Angiography before surgery
  Interventions: Device: CT angiography（CTA）
- Non-CTA Group (No Intervention): The CTA group was routinely peformed upper abdomen enhenced without CT Angiography before surgery

INTERVENTIONS:
Device: CT angiography（CTA） — The CTA group was peformed upper abdomen enhenced and CT Angiography before surgery
  Arms: CTA Group

SUMMARY:
Gastric cancer is one of the most common malignace worldwide, which caused a dramatically death rate, especially in east Asian, such as Japan , South Korea and China. Although the treatment of gastric cancer has a large improvement, such as radiotherapy, chemotherapy and immunotherapy, surgery is yet the mainstream method for the curable malignace without distant metastasis. As the innovation of treatment in gastric caner, laprascopic has gain its popularity owing to its equivalent oncologic outcomes, earlier oral feeding, shorten postopertative of hospital length,compared with open surgery. Depite it has several advantages, the defect of laparascopic surgery is still obvious, such as 2D surgical field, lack of inverse haptic feedback, Inflexible equipment.

D2 Lymph node dissection associated with laparascopic gastronomy is still regard as standard surgical procedure for the gastric cancer patient whose tumor stage was evaluated in advance stage. As we known that the distribution of lymph nod is accompanied with blood vessels, even for well-trained surgeon, the procedure lymph node dissection is a challenging and tough work. Computed Tomography Angiography(3D-CTA), as a emerging technology, is gradually receive the surgeon's attention for its remedy characteristic to the defect of laparascopic surgery, which can visually display the distribution and type of perigastric artery, resulting in decresing the difficulty and risk of surgery.

The aim of the study is to investigate the clinincal outcomes for the patient with BMI ≥25 kg/㎡who underwent laparascopic or robotic gastronomy using CTA to evaluate the type of perigastric artery.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of gastric adenocarcinoma by gastroscopy
2. Age 18~75 years old
3. BMI≥25.0kg/m2
4. Preoperative imaging staging is T1~T4a, N0~3, M0
5. The surgical approach is laparoscopic surgery and robotic surgery

Exclusion Criteria:

1. Patients whose tumors stage are found to be T4b or M1 during the operation, tumors are unresectable and accompanied with malignant tumors in other parts;
2. suffering from other malignant tumors, tumors of low malignant potential (giant cell tumor of bone, pseudomyxadenoma of appendix, invasive fibroma) in the past;
3. Patients who have serious other system diseases and cannot tolerate surgery;
4. Patients with non-adenocarcinoma type malignant tumors in pathology after surgery;
5. Patients with residual gastric cancer;
6. Those who are allergic to iodine contrast agents;
7. Those who have received neoadjuvant therapy before surgery;
8. Pregnant patients;
9. Patients who are participating in other clinical studies trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | during the surgery
  haemorrhagia amount during the operation

SECONDARY OUTCOMES:
Number of lymph node dissection guided by vessel | during the surgery
  the harvest of lymph node during the gastronomy
The total incidence of postoperative complications | 30 days
  the postoperative complications was defined as the complications related to the surgery or systematic,such as pneumonia,urinary tract infection
Postoperative recovery course | 30 days
  Time to first ambulation, flatus, liquid diet and so on
30-day mortality | 30 days
  the 30-day mortality was defined as the death occurs related to the surgery or other occasions within 30 days
hospitalization costs length of hospitalization days | during the hospitalization
  the total cost of hospitalization related to any therapy
3 years OS | 3 years
  3 years overall survival after surgery
3 years DFS | 3 years
  3 years disease free survival after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Yanbing, MD, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Department of Gastrointestinal Surgery, Qingdao University Affiliated Hospital, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Derived] Meng C, Cao S, Li L, Xia L, Chu X, Jiang L, Wang X, Wang H, Huang S, Duan Q, Sun Z, He Q, Hui X, Yang D, Zhang H, Li Z, Liu X, Tian Y, Sun Y, Li Y, Jiang H, Niu Z, Zhang J, Zhou Y. Short-term outcomes of preoperative computed tomography angiography versus standard assessment in patients with BMI >/= 25.0 kg/m2 undergoing laparoscopic gastrectomy: the GISSG20-01 randomized clinical trial. Gastric Cancer. 2025 Mar;28(2):283-293. doi: 10.1007/s10120-024-01580-9. Epub 2025 Jan 9. PMID 39786664
- [Derived] Meng C, Cao S, Liu X, Li L, He Q, Xia L, Jiang L, Chu X, Wang X, Wang H, Hui X, Sun Z, Huang S, Duan Q, Yang D, Zhang H, Tian Y, Li Z, Zhou Y. Effect of preoperative CT angiography examination on the clinical outcome of patients with BMI >/= 25.0 kg/m2 undergoing laparoscopic gastrectomy: study protocol for a multicentre randomized controlled trial. Trials. 2021 Dec 11;22(1):912. doi: 10.1186/s13063-021-05887-1. PMID 34895320